CLINICAL TRIAL: NCT02095145
Title: A Phase IIA Exploratory, Randomized, Placebo-Controlled Trial of Pomegranate Fruit Extract/Pomx™ in Subjects With Clinically Localized Prostate Cancer Undergoing Active Surveillance
Brief Title: Pomegranate-Extract Pill in Preventing Tumor Growth in Patients With Localized Prostate Cancer Undergoing Active Surveillance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2014-00695; NCI-2014-00695 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00033; CO11378 (Other: University of Wisconsin Hospital and Clinics); UWI2013-00-01 (Other: DCP); N01CN00033 (NIH); N01CN35153 (NIH); P30CA014520 (NIH)
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: PSA Level Less Than or Equal to Fifteen; PSA Level Less Than Ten; Stage I Prostate Cancer AJCC v7; Stage II Prostate Cancer AJCC v7; Stage IIA Prostate Cancer AJCC v7; Stage IIB Prostate Cancer AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (pomegranate-extract pill) (Experimental): Patients receive pomegranate-extract pill PO QD for 52 weeks (+/- 1 week).
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Pomegranate-Extract Pill
- Group II (placebo) (Placebo Comparator): Patients receive placebo PO QD for 52 weeks (+/- 1 week).
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Group II (placebo)
Drug: Pomegranate-Extract Pill — Given PO
  Other Names: POMx
  Arms: Group I (pomegranate-extract pill)

SUMMARY:
This randomized phase II trial studies pomegranate-extract pill in preventing tumor growth in patients with prostate cancer that is limited to a certain part of the body (localized), who have chosen observation as their treatment plan. The use of pomegranate-extract pill may slow disease progression in patients with localized prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of pomegranate fruit extract (PFE) 1000 mg, taken daily for 1 year, on the plasma levels of insulin-like growth factor (IGF-1) from baseline to end of study (52 weeks) in participants undergoing active surveillance (AS) for early stage prostate cancer.

SECONDARY OBJECTIVES:

I. To assess compliance with a once daily oral administration of PFE versus placebo over a 52-week period of time.

II. To assess the toxicity of PFE vs. placebo when taken daily for 52 weeks (+/- 1 week).

III. To compare and correlate the effect of 52 weeks of daily dosing with PFE vs placebo on the end of study biopsy results including the presence or absence of tumor, the extent of tumor and Gleason scores.

IV. To compare and correlate the modulation of the following biomarkers with response to PFE versus placebo in three areas of interest: tissue from a completely benign biopsy core, tumor tissue from a positive core, and normal tissue adjacent to tumor from a positive core; plasma: insulin-like growth factor 1/IGF binding protein 3 ratio (IGF-1/IGFBP-3 ratio); prostate tissue (normal and abnormal): apoptosis (CASPASE 3), Ki-67, 8OHdG, IGF-1R, androgen receptor, IGF-1, IGFBP-3, prostate specific antigen (PSA).

V. Measure PFE constituents/metabolites in plasma and urine for evidence of accumulation (trough levels): ellagic acid, dimethyl ellagic acid, dimethyl ellagic acid glucuronide (DMEAG), urolithin A, urolithin A-glucuronide, urolithin B and urolithin B-glucuronide.

VI. Measure PSA doubling time (PSA DT) in serum, using the calculation provided on the Memorial Sloan Kettering Cancer Center website.

VII. To assess the feasibility of cancer chemoprevention trials in a population of men undergoing active surveillance for prostate cancer.

VIII. Measurement of serum testosterone.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive pomegranate-extract pill orally (PO) once daily (QD) for 52 weeks (+/- 1 week).

GROUP II: Patients receive placebo PO QD for 52 weeks (+/- 1 week).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have had a standard-of-care biopsy within 13 months of the baseline study visit and must have been diagnosed with low-grade, clinically localized prostate cancer (Gleason score =< 3+3 with a PSA at baseline < 10 ng/ml in participants < 70 years of age, OR Gleason score =< 3+4 with a PSA at baseline =< 15 ng/ml in participants >= 70 years of age); eligible participants will be those men who are able and willing to undergo AS with PSA monitoring and a scheduled biopsy performed at the end of the study
* No concurrent treatment (hormonal, radiation or systemic chemotherapy) for prostate cancer during study enrollment is planned (unless participants demonstrate clinical evidence of prostate cancer progression such as symptoms, physical exam findings, a rapidly increasing PSA, or radiologic findings which confirm disease progression)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* White blood cells (WBC) >= 3000/mm^3
* Platelets >= 100,000 mm^3
* Hemoglobin >= 10 g/dL
* Total bilirubin =< 1.5 x upper limit of institutional normal
* Alkaline phosphatase =< 1.5 x upper limit of institutional normal
* Aspartate aminotransferase (AST) =< 1.5 x upper limit of institutional normal
* Alanine aminotransferase (ALT) =< 1.5 x upper limit of institutional normal
* Serum creatinine within 1.5 x upper limit of institutional normal
* Sodium 135-144 mmol/L (inclusive)
* Potassium 3.2-4.8 mmol/L (inclusive)
* Participants will be required to use a medically-approved method of birth control or abstinence if their sexual partner is of child-bearing potential
* Participants must be willing to forego foods, beverages and supplements containing pomegranate for the duration of the study
* Ability to understand, and the willingness to sign, a written informed consent document

Exclusion Criteria:

* Any prior surgery to the prostate within 30 days of baseline procedures; NOTE: Biopsies are not considered surgeries
* Evidence of other cancer(s) (excluding non-melanoma skin cancer) within last 5 years
* Prior pelvic radiation for any reason
* Participants cannot be taking 5-alpha-reductase inhibitors while on study or within 6 months of the baseline study visit
* Participants may not be taking carbamazepine (tegretol)
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PFE
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Any significant cardiac event(s) within the 12 months prior to registration, such as episode(s) of symptomatic congestive heart failure, myocardial infarction, unstable angina pectoris or persistent, stable angina pectoris, or cardiac arrhythmia requiring medication

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-05-08 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Jarrard, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Urology San Antonio Research PA, San Antonio, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 38 participants consented, only 30 eligible to start study
Groups:
- Group I (Pomegranate-extract Pill): Patients receive pomegranate-extract pill orally once a day for 52 weeks (+/- 1 week).
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Pomegranate-Extract Pill: Given PO
- Group II (Placebo): Patients receive placebo orally once a day for 52 weeks (+/- 1 week).
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Placebo: Given PO
Period: Overall Study
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo) | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Customized [Count of Participants; unit: Participants]
  Participant Age: 18-64 years | 6 | 8 | 14
  Participant Age: 65 years or older | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants] — The final report for this study contains data for participant 'gender', the study team would like to note this for consistency.
  Participants
    Female | 0 | 0 | 0
    Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 13 | 15 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 15 | 29
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) 0 = Fully active, able to carry on all pre-disease performance without restriction
  1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    ECOG 0 | 14 | 15 | 29
    ECOG 1 | 0 | 0 | 0
Systolic Blood Pressure [Mean (Full Range); unit: mmHg] | 140.71 [115.00 to 162.00] | 139.80 [116.00 to 179.00] | 140.24 [115.00 to 179.00]
Diastolic Blood Pressure [Mean (Full Range); unit: mmHg] | 81.64 [73.00 to 95.00] | 83.60 [71.00 to 108.00] | 82.66 [71.00 to 108.00]
Temperature [Mean (Full Range); unit: degrees Fahrenheit] | 97.81 [96.06 to 98.96] | 97.62 [96.90 to 98.40] | 97.71 [96.06 to 98.96]
Pulse [Mean (Full Range); unit: beats per minute] | 75.00 [55.00 to 91.00] | 68.13 [52.00 to 87.00] | 71.45 [52.00 to 91.00]
Height [Mean (Full Range); unit: cm] | 174.73 [162.56 to 190.50] | 177.23 [160.02 to 188.00] | 176.02 [160.02 to 190.50]
Weight [Mean (Full Range); unit: kg] | 88.92 [67.59 to 102.40] | 94.53 [67.20 to 124.74] | 91.82 [67.20 to 124.74]
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 29.15 [23.12 to 33.53] | 29.91 [25.33 to 35.31] | 29.55 [23.12 to 35.31]
History or Baseline Presence of Disease / Abnormality [Number; unit: participants]
  Skin | 1 | 2 | 3
  Prostate | 2 | 0 | 2
  Head/Eyes/Ears/Neck/Throat | 0 | 1 | 1
  Neurological | 1 | 0 | 1
  Abdomen | 0 | 1 | 1
  Genitalia | 0 | 1 | 1
Gleason Score [Number; unit: scores on a scale] — The Gleason Score is a grading system used to determine the aggressiveness of prostate cancer, scored 1-5 with 1 being healthy tissue and 5 being abnormal. Prostate cancers are assigned 2 scores to define the 2 most prevalent tissue types. They are added together (total range of 2-10). Typical scores fall between 6-10, the higher the overall score, the more likely the cancer will spread.
  scores on a scale
    3+3=6 | 13 | 15 | 28
    3+4=7 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma IGF-1 From Baseline to Post-Treatment
Description: The primary endpoint for modulation of intermediate endpoint biomarkers will be the change in the plasma levels of IGF-1 by a quantitative assay (ELISA) from pre-study to post-treatment. The difference between these time points for the placebo group and the pomegranate fruit extract (PFE) group will be tested using a two-sample t-test with normalizing transformation if necessary or Wilcoxon rank-sum test.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
ng/mL | 19.12 (21.22) | 8.54 (23.11)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Test type: Other; p = 0.190, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Test type: Other; p = 0.211, t-test, 2 sided

2. Secondary Outcome: Compliance: Number of Participants Who Took Study Drug Per Protocol
Description: Summarized by treatment arm with descriptive statistics, and tested for imbalance using Wilcoxon rank-sum test. Reported for each visit per protocol at Week 13, Week 26, Week 39, and Week 52 (end of study).
Time Frame: Up to 1 year
Population: One participant has no compliance values for weeks 26 and 39.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
Participants
  Week 13 | 14 | 14
  Week 26: number analyzed (Participants) | 14 | 14
  Week 26 | 14 | 14
  Week 39: number analyzed (Participants) | 14 | 14
  Week 39 | 14 | 14
  End of Study (Week 52) | 14 | 15

3. Secondary Outcome: Incidence of Adverse Events Graded Per Common Terminology Criteria for Adverse Events (CTCAE)
Description: Patient toxicity throughout the study will be summarized in several ways; the presence or absence of any toxicity, worst CTCAE grade, and strongest investigator-defined relationship will all be examined and characterized by treatment arm, and analyzed appropriately (Wilcoxon rank-sum for ordinal data, Fisher's exact test for dichotomous data, and log rank test for time to event data).
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
Participants
  Any Adverse Event | 14 | 13
  Multiple Adverse Events | 14 | 11
  Grade 3 (Severe) or Worse | 3 | 4
  Serious Adverse Events | 2 | 2

4. Secondary Outcome: Change in Plasma Biomarker Levels From Baseline: IGFBP-3
Description: Differences between the groups will be examined for the change from baseline with the appropriate tests; for dichotomous data Fisher's exact test will be used, for ordinal data Wilcoxon rank-sum test will be used, and for continuous data, and a two-sample t-test with normalizing transformation if necessary or Wilcoxon rank-sum test will be used.
Time Frame: Week 13, Week 26, Week 39, Week 52
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
ng/mL
  Change Baseline to Week 13 | -102.91 (501.07) | -195.57 (592.17)
  Change Baseline to Week 26 | 10.55 (560.69) | 99.74 (652.11)
  Change Baseline to Week 39 | -309.11 (455.91) | 89.34 (381.47)
  Change Baseline to Week 52 | -137.67 (363.48) | -0.39 (498.02)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Baseline to Week 13 p-value; Test type: Other; p = 0.948, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Baseline to Week 26 p-value; Test type: Other; p = 0.711, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Baseline to Week 39 p-value; Test type: Other; p = 0.038, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Baseline to Week 52 p-value; Test type: Other; p = 0.445, Wilcoxon rank-sum test

5. Secondary Outcome: Change in Plasma Biomarker Levels From Baseline: IGF-1/GFBP-3
Description: as for outcome 4
Time Frame: Week 13, Week 26, Week 39, Week 52
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
ratio
  Change Baseline to Week 13 | 0.00 (0.01) | 0.01 (0.01)
  Change Baseline to Week 26 | 0.00 (0.01) | -0.00 (0.01)
  Change Baseline to Week 39 | 0.01 (0.01) | -0.00 (0.01)
  Change Baseline to Week 52 | 0.01 (0.01) | 0.00 (0.01)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Baseline to Week 13 p-value; Test type: Other; p = 0.743, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Baseline to Week 26 p-value; Test type: Other; p = 0.305, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Baseline to Week 39 p-value; Test type: Other; p = 0.111, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Baseline to Week 52 p-value; Test type: Other; p = 0.395, Wilcoxon rank-sum test

6. Secondary Outcome: Change in Total Serum Prostate Specific Antigen (PSA) From Baseline
Time Frame: Up to 1 year
Population: Statistician notes that serum PSA data is missing for one participant in the pomegranate extract arm for all time points, missing for another in the pomegranate arm at week 39, and one from the placebo arm at week 39.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
ng/mL
  Change Baseline to Week 13 | -1.88 (4.78) | -1.05 (1.67)
  Change from Baseline Week 26 | -1.41 (4.67) | -0.77 (1.33)
  Change from Baseline Week 39: number analyzed (Participants) | 14 | 14
  Change from Baseline Week 39 | -1.52 (5.52) | -0.29 (1.91)
  Change Baseline to Week 52 | -1.00 (5.89) | -0.08 (1.83)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline PSA to Week 13; Test type: Other; p = 0.743, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline PSA to Week 26; Test type: Other; p = 0.527, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline PSA to Week 39; Test type: Other; p = 0.879, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline PSA to Week 52; Test type: Other; p = 0.810, Wilcoxon rank-sum test

7. Secondary Outcome: Change in Serum Testosterone
Time Frame: up to 1 year
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
pg/ml
  Baseline | 9.37 (5.23) | 9.73 (3.03)
  Week 26 | 11.43 (10.48) | 12.61 (13.46)
  Week 52 | 14.83 (19.84) | 9.27 (3.42)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Comparison of both arms at baseline; Test type: Other; p = 0.556, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); comparison of both arms at Week 26; Test type: Other; p = 0.647, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); comparison of both arms at end of study, week 52; Test type: Other; p = 0.948, Wilcoxon rank-sum test

8. Secondary Outcome: Prostate Specific Antigen Doubling Time (PSA DT)
Description: PSA DT will be determined from PSA values obtained during study participation (baseline and weeks 13, 26, 39 and 52). The secondary endpoint of PSA DT is based on the value at study completion (week 52 or at point of early termination). However, PSA DT will be determined starting at week 26 (the earliest time point with 3 values) and week 39 and recorded. PSA doubling time is a measure based on the slope of the PSA at multiple time points. If the slope is relatively flat, the predicted doubling time could be far beyond the length of the actual study. As such, the value is not limited to the time frame over which data is collected from the participant.
Time Frame: up to 52 Weeks
Population: One of the participant's PSA values were 'non-detectable', therefore PSA observations could not be calculated for that participant.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 13 | 15
weeks | 134.01 (560.33) | 125.63 (282.90)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Test type: Other; p = 0.580, Wilcoxon rank-sum test

9. Secondary Outcome: Change in Tissue Biomarker Levels: PSA
Description: Compare and correlate biomarker modulation in response to PFE versus placebo in three areas of interest: tissue from a completely benign biopsy core ("benign" in results), tumor tissue from a positive core ("tumor" in results), and normal tissue adjacent to tumor from a positive core ("adjacent" in results). Differences between the groups will be examined for the change from baseline with the appropriate tests; for dichotomous data Fisher's exact test will be used, for ordinal data Wilcoxon rank-sum test will be used, and for continuous data, and a two-sample t-test with normalizing transformation if necessary or Wilcoxon rank-sum test will be used.
Time Frame: Baseline to Week 52
Population: The number analyzed depends on the identification and recovery of relevant tissue type (benign, adjacent, tumor).
Measure: Mean (Standard Deviation); unit: normalized optical density
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
normalized optical density
  Change From Baseline: Benign: number analyzed (Participants) | 13 | 14
  Change From Baseline: Benign | 0.01 (0.42) | 0.04 (0.21)
  Change From Baseline: Adjacent: number analyzed (Participants) | 3 | 5
  Change From Baseline: Adjacent | -0.10 (0.09) | 0.16 (0.43)
  Change From Baseline: Tumor: number analyzed (Participants) | 3 | 5
  Change From Baseline: Tumor | 0.09 (0.39) | 0.25 (0.52)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Benign core p-value; Test type: Other; p = 0.344, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Adjacent core p-value; Test type: Other; p = 0.371, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Tumor core p-value; Test type: Other; p = 0.766, Wilcoxon rank-sum test

10. Secondary Outcome: Change in Tissue Biomarker Levels: IGF-1
Description: Compare and correlate biomarker modulation in response to PFE versus placebo in three areas of interest: tissue from a completely benign biopsy core ("benign" in results), tumor tissue from a positive core ("tumor" in results), and normal tissue adjacent to tumor from a positive core ("adjacent" in results). Measurements for each are per nuclear ("Nuc" in results), cytoplasmic ("Cyt" in results), and cellular ("Cell" in results) basis. Differences between the groups will be examined for the change from baseline with the appropriate tests; for dichotomous data Fisher's exact test will be used, for ordinal data Wilcoxon rank-sum test will be used, and for continuous data, and a two-sample t-test with normalizing transformation if necessary or Wilcoxon rank-sum test will be used.
Time Frame: Baseline to Week 52
Population: The number analyzed depends on the identification and recovery of relevant tissue type (benign, adjacent, tumor).
Measure: Mean (Standard Deviation); unit: normalized optical density
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
normalized optical density
  Change From Baseline: Nuc Benign: number analyzed (Participants) | 12 | 14
  Change From Baseline: Nuc Benign | -0.10 (1.65) | 0.57 (1.91)
  Change From Baseline: Nuc Adjacent: number analyzed (Participants) | 6 | 6
  Change From Baseline: Nuc Adjacent | -0.58 (2.78) | 1.74 (1.45)
  Change From Baseline: Nuc Tumor: number analyzed (Participants) | 6 | 6
  Change From Baseline: Nuc Tumor | -0.53 (2.39) | 1.06 (1.41)
  Change From Baseline: Cyt Benign: number analyzed (Participants) | 12 | 14
  Change From Baseline: Cyt Benign | -0.43 (1.35) | 0.21 (1.38)
  Change From Baseline: Cyt Adjacent: number analyzed (Participants) | 6 | 6
  Change From Baseline: Cyt Adjacent | -0.52 (1.77) | 1.47 (1.15)
  Change From Baseline: Cyt Tumor: number analyzed (Participants) | 6 | 6
  Change From Baseline: Cyt Tumor | -0.65 (1.64) | 1.10 (1.01)
  Change From Baseline: Cell Benign: number analyzed (Participants) | 12 | 14
  Change From Baseline: Cell Benign | -0.29 (1.45) | 0.35 (1.58)
  Change From Baseline: Cell Adjacent: number analyzed (Participants) | 6 | 6
  Change From Baseline: Cell Adjacent | -0.53 (2.17) | 1.59 (1.18)
  Change From Baseline: Cell Tumor: number analyzed (Participants) | 6 | 6
  Change From Baseline: Cell Tumor | -0.61 (1.99) | 1.06 (1.02)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: IGF-1 Benign (Nuc); Test type: Other; p = 0.304, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: IGF-1 Adjacent (Nuc); Test type: Other; p = 0.230, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: IGF-1 Tumor (Nuc); Test type: Other; p = 0.298, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: IGF-1 Benign (Cyt); Test type: Other; p = 0.247, Wilcoxon rank-sum test
Statistical Analysis 5: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: IGF-1 Adjacent (Cyt); Test type: Other; p = 0.093, Wilcoxon rank-sum test
Statistical Analysis 6: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: IGF-1 Tumor (Cyt); Test type: Other; p = 0.066, Wilcoxon rank-sum test
Statistical Analysis 7: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: IGF-1 Benign (Cell); Test type: Other; p = 0.247, Wilcoxon rank-sum test
Statistical Analysis 8: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: IGF-1 Adjacent (Cell); Test type: Other; p = 0.128, Wilcoxon rank-sum test
Statistical Analysis 9: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: IGF-1 Tumor (Cell); Test type: Other; p = 0.128, Wilcoxon rank-sum test

11. Secondary Outcome: Change in Tissue Biomarker Levels: IGFBP-3
Description: as for outcome 10
Time Frame: Baseline to Week 52
Population: The number analyzed depends on the identification and recovery of relevant tissue type (benign, adjacent, tumor).
Measure: Mean (Standard Deviation); unit: normalized optical density
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
normalized optical density
  Change From Baseline: Nuc Benign: number analyzed (Participants) | 13 | 14
  Change From Baseline: Nuc Benign | -0.43 (2.77) | 0.78 (3.70)
  Change From Baseline: Nuc Adjacent: number analyzed (Participants) | 3 | 5
  Change From Baseline: Nuc Adjacent | 0.01 (1.51) | 1.55 (1.90)
  Change From Baseline: Nuc Tumor: number analyzed (Participants) | 3 | 5
  Change From Baseline: Nuc Tumor | 0.69 (2.21) | 1.75 (1.79)
  Change From Baseline: Cyt Benign: number analyzed (Participants) | 13 | 14
  Change From Baseline: Cyt Benign | -0.38 (1.56) | 0.52 (1.26)
  Change From Baseline: Cyt Adjacent: number analyzed (Participants) | 3 | 5
  Change From Baseline: Cyt Adjacent | -0.96 (1.39) | 0.67 (0.90)
  Change From Baseline: Cyt Tumor: number analyzed (Participants) | 3 | 5
  Change From Baseline: Cyt Tumor | -1.09 (0.90) | 0.76 (0.80)
  Change From Baseline: Cell Benign: number analyzed (Participants) | 13 | 14
  Change From Baseline: Cell Benign | -0.43 (2.02) | 0.68 (2.39)
  Change From Baseline: Cell Adjacent: number analyzed (Participants) | 3 | 5
  Change From Baseline: Cell Adjacent | -0.24 (1.62) | 1.07 (1.13)
  Change From Baseline: Cell Tumor: number analyzed (Participants) | 3 | 5
  Change From Baseline: Cell Tumor | -0.14 (1.48) | 1.24 (0.79)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Nuc Benign p-value; Test type: Other; p = 0.297, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Nuc Adjacent p-value; Test type: Other; p = 0.233, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Nuc Tumor p-value; Test type: Other; p = 0.371, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cyt Benign p-value; Test type: Other; p = 0.198, Wilcoxon rank-sum test
Statistical Analysis 5: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cyt Adjacent p-value; Test type: Other; p = 0.233, Wilcoxon rank-sum test
Statistical Analysis 6: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cyt Tumor p-value; Test type: Other; p = 0.074, Wilcoxon rank-sum test
Statistical Analysis 7: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cell Benign p-value; Test type: Other; p = 0.234, Wilcoxon rank-sum test
Statistical Analysis 8: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cell Adjacent p-value; Test type: Other; p = 0.233, Wilcoxon rank-sum test
Statistical Analysis 9: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cell Tumor p-value; Test type: Other; p = 0.233, Wilcoxon rank-sum test

12. Secondary Outcome: Change in Tissue Biomarker Levels: CASP3
Description: as for outcome 10
Time Frame: Baseline to Week 52
Population: The number analyzed depends on the identification and recovery of relevant tissue type (benign, adjacent, tumor).
Measure: Mean (Standard Deviation); unit: normalized optical density
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
normalized optical density
  Change From Baseline: Nuc Benign: number analyzed (Participants) | 13 | 14
  Change From Baseline: Nuc Benign | -0.61 (1.74) | 0.57 (1.74)
  Change From Baseline: Nuc Adjacent: number analyzed (Participants) | 4 | 5
  Change From Baseline: Nuc Adjacent | -0.40 (1.06) | 0.38 (1.55)
  Change From Baseline: Nuc Tumor: number analyzed (Participants) | 4 | 5
  Change From Baseline: Nuc Tumor | -0.34 (1.06) | 0.04 (0.43)
  Change From Baseline: Cyt Benign: number analyzed (Participants) | 13 | 14
  Change From Baseline: Cyt Benign | -0.49 (1.43) | -0.01 (1.30)
  Change From Baseline: Cyt Adjacent: number analyzed (Participants) | 4 | 5
  Change From Baseline: Cyt Adjacent | -0.42 (1.31) | 0.54 (1.44)
  Change From Baseline: Cyt Tumor: number analyzed (Participants) | 4 | 5
  Change From Baseline: Cyt Tumor | -0.45 (1.66) | -0.00 (0.33)
  Change From Baseline: Cell Benign: number analyzed (Participants) | 13 | 14
  Change From Baseline: Cell Benign | -0.54 (1.52) | 0.23 (1.40)
  Change From Baseline: Cell Adjacent: number analyzed (Participants) | 4 | 5
  Change From Baseline: Cell Adjacent | -0.40 (1.16) | 0.43 (1.42)
  Change From Baseline: Cell Tumor: number analyzed (Participants) | 4 | 5
  Change From Baseline: Cell Tumor | -0.35 (1.35) | 0.01 (0.36)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Nuc Benign p-value; Test type: Other; p = 0.167, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Nuc Adjacent p-value; Test type: Other; p = 0.391, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Nuc Tumor p-value; Test type: Other; p = 0.713, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cyt Benign p-value; Test type: Other; p = 0.452, Wilcoxon rank-sum test
Statistical Analysis 5: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cyt Adjacent p-value; Test type: Other; p = 0.391, Wilcoxon rank-sum test
Statistical Analysis 6: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cyt Tumor p-value; Test type: Other; p = 0.713, Wilcoxon rank-sum test
Statistical Analysis 7: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cell Benign p-value; Test type: Other; p = 0.344, Wilcoxon rank-sum test
Statistical Analysis 8: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cell Adjacent p-value; Test type: Other; p = 0.391, Wilcoxon rank-sum test
Statistical Analysis 9: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cell Tumor p-value; Test type: Other; p = 0.713, Wilcoxon rank-sum test

13. Secondary Outcome: Change in Tissue Biomarker Levels: Ki-67
Description: as for outcome 9
Time Frame: Baseline to Week 52
Population: The number analyzed depends on the identification and recovery of relevant tissue type (benign, adjacent, tumor).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
percent change
  Change From Baseline: Benign: number analyzed (Participants) | 13 | 14
  Change From Baseline: Benign | 0.01 (0.50) | 0.06 (0.52)
  Change From Baseline: Adjacent: number analyzed (Participants) | 4 | 5
  Change From Baseline: Adjacent | -0.27 (0.36) | -0.53 (1.73)
  Change From Baseline:Tumor: number analyzed (Participants) | 4 | 5
  Change From Baseline:Tumor | -6.40 (12.11) | 1.31 (0.89)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Benign p-value; Test type: Other; p = 0.865, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Adjacent p-value; Test type: Other; p = 1.000, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Tumor p-value; Test type: Other; p = 0.066, Wilcoxon rank-sum test

14. Secondary Outcome: Change in Tissue Biomarker Levels: IGF-Rb
Description: as for outcome 10
Time Frame: Baseline to Week 52
Population: The number analyzed depends on the identification and recovery of relevant tissue type (benign, adjacent, tumor).
Measure: Mean (Standard Deviation); unit: normalized optical density
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
normalized optical density
  Change From Baseline: Nuc Benign: number analyzed (Participants) | 12 | 14
  Change From Baseline: Nuc Benign | -0.50 (1.08) | -0.52 (1.03)
  Change From Baseline: Nuc Adjacent: number analyzed (Participants) | 4 | 5
  Change From Baseline: Nuc Adjacent | 0.62 (1.24) | 0.32 (0.37)
  Change From Baseline: Nuc Tumor: number analyzed (Participants) | 4 | 5
  Change From Baseline: Nuc Tumor | 0.63 (2.00) | 0.88 (0.50)
  Change From Baseline: Cyt Benign: number analyzed (Participants) | 12 | 14
  Change From Baseline: Cyt Benign | 0.09 (1.35) | -0.48 (1.19)
  Change From Baseline: Cyt Adjacent: number analyzed (Participants) | 4 | 5
  Change From Baseline: Cyt Adjacent | -0.24 (0.71) | 0.80 (0.94)
  Change From Baseline: Cyt Tumor: number analyzed (Participants) | 4 | 5
  Change From Baseline: Cyt Tumor | 0.04 (1.45) | 0.58 (0.42)
  Change From Baseline: Cell Benign: number analyzed (Participants) | 12 | 14
  Change From Baseline: Cell Benign | -0.19 (1.21) | -0.52 (1.05)
  Change From Baseline: Cell Adjacent: number analyzed (Participants) | 4 | 5
  Change From Baseline: Cell Adjacent | 0.17 (0.85) | 0.56 (0.52)
  Change From Baseline: Cell Tumor: number analyzed (Participants) | 4 | 5
  Change From Baseline: Cell Tumor | 0.31 (1.63) | 0.73 (0.39)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Nuc Benign p-value; Test type: Other; p = 1.000, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Nuc Adjacent p-value; Test type: Other; p = 0.903, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Nuc Tumor p-value; Test type: Other; p = 1.000, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Cyt Benign p-value; Test type: Other; p = 0.269, Wilcoxon rank-sum test
Statistical Analysis 5: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Cyt Adjacent p-value; Test type: Other; p = 0.066, Wilcoxon rank-sum test
Statistical Analysis 6: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Cyt Tumor p-value; Test type: Other; p = 1.000, Wilcoxon rank-sum test
Statistical Analysis 7: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Cell Benign p-value; Test type: Other; p = 0.425, Wilcoxon rank-sum test
Statistical Analysis 8: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Cell Adjacent p-value; Test type: Other; p = 0.270, Wilcoxon rank-sum test
Statistical Analysis 9: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Cell Tumor p-value; Test type: Other; p = 1.000, Wilcoxon rank-sum test

15. Secondary Outcome: Change in Tissue Biomarker Levels: 8OHdG
Description: as for outcome 10
Time Frame: Baseline to Week 52
Population: The number analyzed depends on the identification and recovery of relevant tissue type (benign, adjacent, tumor).
Measure: Mean (Standard Deviation); unit: normalized optical density
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
normalized optical density
  Change From Baseline: Nuc Benign: number analyzed (Participants) | 12 | 14
  Change From Baseline: Nuc Benign | -0.05 (0.15) | -0.02 (0.15)
  Change From Baseline: Nuc Adjacent: number analyzed (Participants) | 6 | 6
  Change From Baseline: Nuc Adjacent | -0.09 (0.13) | 0.07 (0.16)
  Change From Baseline: Nuc Tumor: number analyzed (Participants) | 6 | 6
  Change From Baseline: Nuc Tumor | -0.15 (0.08) | 0.07 (0.20)
  Change From Baseline: Cyt Benign: number analyzed (Participants) | 12 | 14
  Change From Baseline: Cyt Benign | -0.15 (0.47) | 0.21 (0.54)
  Change From Baseline: Cyt Adjacent: number analyzed (Participants) | 6 | 6
  Change From Baseline: Cyt Adjacent | -0.28 (0.45) | 0.47 (0.54)
  Change From Baseline: Cyt Tumor: number analyzed (Participants) | 6 | 6
  Change From Baseline: Cyt Tumor | -0.58 (0.33) | 0.41 (0.52)
  Change From Baseline: Cell Benign: number analyzed (Participants) | 12 | 14
  Change From Baseline: Cell Benign | -0.17 (0.43) | 0.09 (0.39)
  Change From Baseline: Cell Adjacent: number analyzed (Participants) | 6 | 6
  Change From Baseline: Cell Adjacent | -0.31 (0.43) | 0.20 (0.40)
  Change From Baseline: Cell Tumor: number analyzed (Participants) | 6 | 6
  Change From Baseline: Cell Tumor | -0.50 (0.28) | 0.19 (0.47)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Nuc Benign p-value; Test type: Other; p = 0.625, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Nuc Adjacent p-value; Test type: Other; p = 0.128, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Nuc Tumor p-value; Test type: Other; p = 0.045, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cyt Benign p-value; Test type: Other; p = 0.105, Wilcoxon rank-sum test
Statistical Analysis 5: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cyt Adjacent p-value; Test type: Other; p = 0.066, Wilcoxon rank-sum test
Statistical Analysis 6: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cyt Tumor p-value; Test type: Other; p = 0.005, Wilcoxon rank-sum test
Statistical Analysis 7: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cell Benign p-value; Test type: Other; p = 0.129, Wilcoxon rank-sum test
Statistical Analysis 8: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cell Adjacent p-value; Test type: Other; p = 0.066, Wilcoxon rank-sum test
Statistical Analysis 9: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change From Baseline: Cell Tumor p-value; Test type: Other; p = 0.013, Wilcoxon rank-sum test

16. Secondary Outcome: Change in Tissue Biomarker Levels: AR
Description: as for outcome 9
Time Frame: Baseline to Week 52
Population: The number analyzed depends on the identification and recovery of relevant tissue type (benign, adjacent, tumor).
Measure: Mean (Standard Deviation); unit: normalized optical density
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
normalized optical density
  Change From Baseline: Benign: number analyzed (Participants) | 12 | 14
  Change From Baseline: Benign | 0.48 (1.07) | -0.55 (1.87)
  Change From Baseline: Adjacent: number analyzed (Participants) | 4 | 5
  Change From Baseline: Adjacent | -0.38 (0.60) | 1.02 (0.90)
  Change From Baseline: Tumor: number analyzed (Participants) | 4 | 5
  Change From Baseline: Tumor | -1.22 (1.15) | 0.38 (0.94)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Benign p-value; Test type: Other; p = 0.143, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Adjacent p-value; Test type: Other; p = 0.037, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline: Tumor p-value; Test type: Other; p = 0.111, Wilcoxon rank-sum test

17. Secondary Outcome: Change in Levels of Pomegranate Fruit Extract (PFE) Constituents/Metabolites: Urolithin A
Description: as for outcome 4
Time Frame: Change from Baseline at Week 13, Week 26, Week 39, and Week 52
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
ng
  Change from Baseline Week 13 | 13491.88 (25612.57) | -8722.87 (32254.35)
  Change from Baseline Week 26 | 29686.34 (38169.43) | -7119.63 (33532.58)
  Change from Baseline Week 39 | 41322.95 (80948.44) | -3688.76 (32749.71)
  Change from Baseline Week 52 | 21622.01 (29672.67) | -4882.23 (17075.55)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline Week 13; Test type: Other; p = 0.068, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline Week 26; Test type: Other; p = 0.004, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline Week 39; Test type: Other; p = 0.002, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline Week 52; Test type: Other; p < 0.001, Wilcoxon rank-sum test

18. Secondary Outcome: Change in Levels of PFE Constituents/Metabolites: Urolithin B
Description: as for outcome 4
Time Frame: Change from Baseline at Week 13, Week 26, Week 39, and Week 52
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
ng
  Change from Baseline Week 13 | 0.00 (0.00) | 0.00 (0.00)
  Change from Baseline Week 26 | 0.00 (0.00) | 156.86 (603.11)
  Change from Baseline Week 39 | 709.24 (2653.74) | 801.40 (2807.45)
  Change from Baseline Week 52 | 1389.82 (4536.11) | 216.54 (838.66)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline Week 13; Test type: Other; p = 1.000, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Pomegranate-extract Pill); Change from Baseline Week 26; Test type: Other; p = 0.180, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline Week 39; Test type: Other; p = 0.620, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change from Baseline Week 52; Test type: Other; p = 0.536, Wilcoxon rank-sum test

19. Secondary Outcome: Change in Gleason Score
Description: The Gleason Score is a grading system used to determine the aggressiveness of prostate cancer, scored 1-5 with 1 being healthy tissue and 5 being abnormal. Prostate cancers are assigned 2 scores to define the 2 most prevalent tissue types. They are added together (total range of 2-10). Typical scores fall between 6-10, the higher the overall score, the more likely the cancer will spread.
Time Frame: Baseline to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 14 | 15
Participants
  Baseline: 0+0=0 | 0 | 0
  Baseline: 3+3=6 | 13 | 15
  Baseline: 3+4=7 | 1 | 0
  Surgery Visit (52 Weeks): 0+0=0 | 5 | 6
  Surgery Visit (52 Weeks): 3+3=6 | 7 | 8
  Surgery Visit (52 Weeks): 3+4=7 | 2 | 1

20. Secondary Outcome: Change in Biopsy Tumor Involvement on Prostate Biopsy
Description: Change in the length of biopsy cores that contained cancerous tissue from Baseline to end of study.
Time Frame: Baseline to 1 year
Population: One participant has a baseline measurement but does not have an end of study measurement, a change in the biopsy tumor involvement for this participant is therefore not possible to calculate.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
Number analyzed (Participants) | 13 | 15
mm | 0.34 (8.09) | 1.88 (8.36)
Statistical Analysis 1: Comparison: Group I (Pomegranate-extract Pill) vs Group II (Placebo); Change in Tumor Volume from baseline to end of study per arm; Test type: Other; p = 0.231, Wilcoxon rank-sum test

ADVERSE EVENTS:
Time Frame: up to 52 weeks
Arm/Group | Group I (Pomegranate-extract Pill) | Group II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/14 | 2/15
Other Adverse Events (participants affected / at risk) | 14/14 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Pomegranate-extract Pill) (N=14) | Group II (Placebo) (N=15)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Surgical and Medical Procedures, other (Surgical and medical procedures) | 1 (1) | 0 (0)
Post-Operative Hemorrhage (Surgical and medical procedures) | 1 (1) | 0 (0)
Abdominal Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Pomegranate-extract Pill) (N=14) | Group II (Placebo) (N=15)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Infections and Infestations, Other (Infections and infestations) | 1 (1) | 0 (0)
Surgical and Medical Procedures (Surgical and medical procedures) | 2 (2) | 4 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cardiac Disorders, other (Cardiac disorders) | 0 (0) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Investigations, other (Investigations) | 1 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Eye Disorders, Other (Eye disorders) | 0 (0) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Blood and Lymphatic System, other (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 10 (18) | 8 (16)
Skin and Subcutaneous Tissue Disorders, Other (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis Noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal and Urinary Disorders, Other (Renal and urinary disorders) | 1 (1) | 1 (2)
Renal Calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Urgency (Renal and urinary disorders) | 1 (1) | 1 (1)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Sinus Pain (Nervous system disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Range of Motion Decreased Lumbar Spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Cholesterol High (Investigations) | 2 (2) | 0 (0)
Creatinine Increased (Investigations) | 1 (1) | 0 (0)
Post-Operative Hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal Infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 1 (1) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 2 (4) | 3 (5)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02095145/Prot_SAP_ICF_000.pdf